CLINICAL TRIAL: NCT05219851
Title: The Risk Factors for Acute Radiation Pneumonitis in Patients With Prior Receipt of Immune Checkpoint Inhibitors.in Real-world Clinical Practice: a Multicenter, Prospective, Open, Non-interventional Study
Brief Title: The Risk Factors for Acute Radiation Pneumonitis in Patients With Prior Receipt of Immune Checkpoint Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, Clinical Professor, Hubei Cancer Hospital
Other Study IDs: HBCH-RT-2022-RP
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cancer Patients
Keywords: IMRT; Radiotherapy; Immune checkpoint inhibitor; Pneumonitis; Risk factors
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Cancer patients underwent thoracic intensity-modulated radiotherapy — Cancer patients underwent thoracic intensity-modulated radiotherapy, previously received ICIs

SUMMARY:
The purpose of this non-interventional study is to collect data on the risk factors for acute radiation pneumonitis in patients with prior receipt of immune checkpoint inhibitors.

DETAILED DESCRIPTION:
1. Incidence of acute radiation pneumonitis (aRPs) in in patients with prior receipt of immune checkpoint inhibitors.
2. Risk factors (especially analysis of the dosimetric risk factor) which may affect the product of aRPs events.
3. Establish a model to predict aRPs and guide clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed malignant tumor
2. Cancer patients with previously received ICIs underwent thoracic intensity-modulated radiotherapy

Exclusion Criteria:

1. Cancer patients did not receive immunotherapy before thoracic intensity-modulated radiotherapy
2. Non-thoracic radiotherapy patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with the product will be enrolled in the investigation
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute radiation pneumonitis (aRPs) in patients with prior receipt of immune checkpoint inhibitors. | 6 months after last-patient- radiation
  All suspected diagnoses of pneumonitis (regardless of grade) were centrally reviewed by a multidisciplinary committee consisting of at least one radiologist, pulmonologist, and oncologist. CT (or PET-CT) imaging was reviewed for each patient, which was then compared to the radiation treatment plan; other causes such as infection or tumor progression had to be ruled out using the appropriate workup.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No